CLINICAL TRIAL: NCT06124456
Title: Vigorous- Versus Moderate-intensity Exercise to Reduce Liver Fat in Adults With Obesity and Non-alcoholic Fatty Liver Disease (NAFLD): A Randomized Controlled Equivalence Trial
Brief Title: Vigorous- Versus Moderate-intensity Exercise to Reduce Liver Fat in Adults With Obesity and NAFLD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Parco M. Siu, PhD, Professor and Division Head, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HKU-NFI
Record Dates: First submitted 2023-11-03; First posted 2023-11-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Obesity; NAFLD
Keywords: NAFLD; Obesity; Liver Fat; exercise
MeSH Terms: conditions — Obesity; Non-alcoholic Fatty Liver Disease; Fatty Liver; Motor Activity

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly allocated to the usual care control or moderate- or vigorous-intensity walking groups on a 1:1:1 basis using block randomization with a block size between 6 and 12. Randomization will be implemented by the biostatistician Co-I or his delegate, who will not interact with the subjects or research personnel during recruitment to avoid allocation bias. The research personnel will then obtain the sequence for each subject to ensure allocation concealment.
Who Masked: Outcomes Assessor
Masking Description: Random allocation will be performed after subjects have completed the baseline assessments. Subjects and the research personnel delivering the walking program and health education cannot be blinded to group allocation, but the latter will not be involved in the outcome assessments. All personnel involved in the outcome assessments will be blinded to the group allocation, and subjects will be instructed not to disclose their allocation during the assessments. The research personnel conducting the statistical analysis cannot be fully blinded to the treatment allocation for the between-group comparisons but will be blinded to subjects' identity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care Control Group (Placebo Comparator)
  Interventions: Other: Usual Care Control Group
- Moderate-intensity Exercise Intervention (Experimental)
  Interventions: Other: Moderate-intensity Exercise Intervention
- Vigorous-intensity Exercise Intervention (Experimental)
  Interventions: Other: Vigorous-intensity Exercise Intervention

INTERVENTIONS:
Other: Usual Care Control Group — Subjects in the usual care control group will receive health education as the attention control. The program will consist of eight 150-minute bi-weekly sessions covering major health issues relating to general health and NAFLD, to be obtained from publicly accessible resources from the Hong Kong Department of Health. Health education information on non-communicable diseases (e.g., cancers, diabetes, coronary heart diseases, obesity, and mental illness), infectious diseases (e.g., COVID-19), and a healthy lifestyle (e.g., balanced diet, physical activity, good sleep, tobacco use, alcohol cessation, and stress management) will also be distributed to the subjects in the exercise groups through recorded presentation videos and leaflets/pamphlets during the first 16 weeks.
  Arms: Usual Care Control Group
Other: Moderate-intensity Exercise Intervention — The walking time in each session will be 50 minutes for the moderate-intensity group. The overall weekly exercise volume for the two groups will be the same based on total energy expenditure, as per the WHO's physical activity recommendation (150 minutes of moderate-intensity physical activity weekly is equivalent to 75 minutes of vigorous-intensity physical activity weekly). Five minutes of walking at a normal pace will be included for warm-up and cool-down.
  Arms: Moderate-intensity Exercise Intervention
Other: Vigorous-intensity Exercise Intervention — The walking time in each session will be 25 minutes for the vigorous-intensity group. The overall weekly exercise volume for the two groups will be the same based on total energy expenditure, as per the WHO's physical activity recommendation (150 minutes of moderate-intensity physical activity weekly is equivalent to 75 minutes of vigorous-intensity physical activity weekly). Five minutes of walking at a normal pace will be included for warm-up and cool-down.
  Arms: Vigorous-intensity Exercise Intervention

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) arising from obesity has become a global health concern. Although exercise is a cornerstone approach for managing NAFLD, detailed exercise prescription guidelines are unavailable. According to World Health Organization (WHO) recommendations, 1 minute of vigorous-intensity physical activity can achieve equivalent health benefits to 2 minutes of moderate-intensity physical activity. It is not known whether this relationship is applicable to exercise prescribed as an adjunct therapy in NAFLD treatment. The answer has public health implications because people living with NAFLD can potentially opt for safe higher-intensity exercise requiring less of a time commitment, whereas those in older age groups or with comorbidities, for whom vigorous exercise is unsuitable, can adopt a moderate-intensity regimen of longer duration to acquire equivalent therapeutic outcomes. Adults with obesity and NAFLD will be randomly allocated to a supervised vigorous- or moderate-intensity walking group or usual care control group. Each exercise group will receive a 16-week intervention comprising three walking sessions weekly, whereas the usual care group will receive general health education as the attention control. The per-session walking time will be 25 minutes for the vigorous group and 50 minutes for the moderate group, equating to the same weekly exercise volume and caloric expenditure for each group according to the WHO's minimum physical activity recommendation. Outcome measures, including liver fat, visceral and body fat, body anthropometry, intervention adherence, psychological measures, health-related quality of life, medication usage, adverse events, habitual physical activity, and diet, will be examined by assessors blinded to the group allocation at baseline, 16 weeks (post-intervention), and 42 weeks (26-week post-intervention follow-up). Data will be analyzed by generalized estimating equations and linear contrasts. The proposed study will provide evidence on the presumed equivalent benefits of vigorous- and moderate-intensity exercise, with a follow-up period allowing assessment of the efficacy, safety, adherence, and sustainability of each. The findings will inform practitioners of the role of exercise intensity in reducing liver fat and refine the exercise guidelines for NAFLD patients.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) arising from obesity has become a global health concern. As well as being a risk factor for cardiovascular disease, diabetes, and chronic kidney disease, it has also been identified as a precursor to severe liver disease. Given that there is no available licensed drug for the treatment of NAFLD, the proposed research seeks to contribute to the treatment and management of NAFLD by comparing two walking exercise regimens as a lifestyle intervention. Using a robust randomized controlled equivalence trial design, it will seek an answer to this research question: Does vigorous-intensity exercise induce equivalent benefits in reducing liver fat relative to moderate-intensity exercise at matched weekly exercise volumes aligned with the World Health Organization's (WHO) minimum physical activity recommendation, and can the two regimens improve NAFLD to a similar degree? Our results are expected to provide scientific evidence-based conclusions revealing the optimal exercise intensity for NAFLD treatment in patients with obesity. The proposed study is novel, with worldwide implications for NAFLD management. The walking programs will be delivered in accordance with the WHO's minimal physical activity recommendations, thereby putting into practice the standardized WHO physical activity guidelines, even for unfit beginners for whom minimal exercise is a more feasible goal. The project thus has two objectives:

1. To examine the therapeutic efficacy of a walking exercise intervention, at either moderate- or vigorous-intensity, for reducing liver fat in adults with obesity and NAFLD. The two exercise intensities to be tested are based on the operational definition of the WHO, and the weekly exercise volumes are aligned with the WHO's minimum physical activity recommendation.

   It is important to elucidate the practical value of the therapeutic efficacy of the walking exercise intervention, at either moderate- or vigorous-intensity, because inactive patients with obesity begin exercise training programs with lower, more achievable goals to learn how to train safely and then adapt progressively, thereby building a sense of self-efficacy and self-confidence to continue adherence. Hence, the proposed research has practical value, as it will provide research evidence on the WHO's minimum exercise guidelines, ultimately contributing to the management and treatment of NAFLD among obese adults.
2. To compare the equivalence of the head-to-head therapeutic efficacy of moderate-intensity exercise versus vigorous-intensity exercise with matched weekly exercise volumes for reducing liver fat in adults with obesity and NAFLD.

This study has important scientific and practical value because it will address an unanswered scientific question: Does vigorous-intensity exercise induce equivalent benefits for reducing liver fat in comparison with moderate-intensity exercise at matched weekly exercise volumes? Its findings will be of practical public health significance to people living with obesity and NAFLD, as they will have the option to engage in vigorous-intensity exercise for a shorter duration or moderate-intensity exercise for a longer duration, following the WHO's physical activity recommendation (75 minutes of vigorous-intensity or 150 minutes of moderate-intensity exercise weekly). This flexibility aligns with the concept of "personalized medicine" and is likely to facilitate patient adherence to an exercise program. If the results show a moderate-intensity exercise regimen with a longer per-session exercise duration to demonstrate an equivalent therapeutic response, the study will also be of important clinical value, especially for patients in older age groups or those with comorbidities, who may be frail and unable to participate in vigorous-intensity exercise. The proposed research is thus expected to provide new evidence to refine the exercise guidelines for NAFLD patients, thereby guiding these patients and their healthcare professionals as to the intensity of weekly exercise that is most suited to their personal circumstances and lifestyles.

The investigators will test two hypotheses: 1) a 16-week moderate- or vigorous-intensity walking intervention, when delivered at the minimum amount of physical activity recommended by the WHO, significantly reduces liver fat in adults with obesity and NAFLD compared with a usual care control group (to be tested through designed superiority comparisons between the moderate/vigorous groups and control group), and 2) the therapeutic efficacy of vigorous-intensity exercise for reducing liver fat is equivalent to that of moderate-intensity exercise at matched weekly exercise volumes (i.e., 75 minutes of vigorous-intensity physical activity versus 150 minutes of moderate-intensity physical activity weekly) (to be tested through designed equivalence comparison between the vigorous and moderate groups).

ELIGIBILITY:
Inclusion Criteria:

* Cantonese, Mandarin, or English-speaking Chinese,
* aged 18-69,
* centrally obese according to the Asia-specific cut-off (waist circumference 90 cm for males, 80 cm for females) and BMI ≥23 (i.e., overweight as defined by the Hong Kong government),
* with NAFLD (defined as >5% intrahepatic triglycerides assessed by 1H-MR spectroscopy),
* able to perform the prescribed exercise program. Both men and women will be included to enhance generalizability.

Exclusion Criteria:

* regular exercise training (>3 sessions of >60 min of moderate-intensity exercise training weekly) in the past 6 months,
* medical history of cardiovascular disease, chronic pulmonary or kidney disease, heart failure, cancer, and/or liver disease except NAFLD,
* somatic conditions that limit exercise participation (e.g., limb loss),
* impaired mobility due to chronic disease (e.g., chronic arthritis/osteoarthritis, neurological, musculoskeletal, and autoimmune diseases),
* daily smoking habit,
* excess alcohol consumption (daily ≥20 g of alcohol for men and ≥10 g for women) in the past 1 year,
* consumption of certain drugs (e.g., tamoxifen and estrogen) known to be secondary causes of steatosis,
* surgery and therapy for morbid obesity in the past 6 months and during the study period (e.g., gastric bypass, gastric band, sleeve gastrectomy, gastric reduction duodenal switch, or dietitian-prescribed dietary program).

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Liver Fat | 16 weeks
  Intrahepatic triglycerides will be examined using 1H-MR spectroscopy in a 3×3×3 cm voxel using a 3.0T system. A trained MRI technician will operate the machine, position the subjects, and analyze the results.

SECONDARY OUTCOMES:
Liver Fat | 42 weeks
  Intrahepatic triglycerides will be examined using 1H-MR spectroscopy in a 3×3×3 cm voxel using a 3.0T system. A trained MRI technician will operate the machine, position the subjects, and analyze the results.
Visceral Adiposity | 16 weeks, 42 weeks
  Abdominal visceral fat will be measured between the thoracic diaphragm and upper border of the first sacral vertebra using a 3.0T system. A trained MRI technician will operate the machine, position the subjects, and analyze the results.
Body Adiposity | 16 weeks, 42 weeks
  Total body fat mass will be determined using a full-body DXA scanner. A trained technician will operate the DXA machine, position the subjects, and analyze the results.
Body Anthropometry-Height | 16 weeks, 42 weeks
  Measuring height in meters (m).
Body Anthropometry- Weight | 16 weeks, 42 weeks
  Measuring weight in kilograms (kg).
Body Anthropometry- BMI | 16 weeks, 42 weeks
  BMI will be determined by the equation BMI (kg/m2) = bodyweight/height^2. A calibrated electronic digital weighing scale with a 200 kg capacity and ± 0.05 kg accuracy will be used to weigh the subjects. A stadiometer with a 200 cm limit and ± 0.01 cm accuracy will be used to measure body height.
Medication | 16 weeks, 42 weeks
  Subjects' use of and detailed information on medications for chronic health conditions will be recorded at baseline. Subjects will be allowed to alter their dosage as advised by their physicians over the study period, which will be recorded as a secondary outcome. Data on medication dose and weekly frequency will be presented as the total lowest recommended dose in 7 days for analysis.
Cardiorespiratory Fitness | 16 weeks, 42 weeks
  The VO2max test will be conducted using a calibrated motor-driven treadmill, continuous metabolic VO2 will be measured using a COSMED Quark CPET gas analysis system, and continuous electrocardiogram will be monitored using a 12-lead wireless COSMED Quark T12x system. The test will be performed using the modified Bruce protocol, which is routinely used by our team. The Borg rate of perceived exertion and heart rate will be continuously recorded. The maximal attainable heart rate is the peak heart rate.
Health-related Quality of Life | 16 weeks, 42 weeks
  The Chronic Liver Disease Questionnaire (CLDQ-NAFLD), a fully validated disease-specific instrument, will be used to measure health-related quality of life. The instrument has 36 items grouped into six domains (abdominal symptoms, activity, emotional, fatigue, systemic symptoms, and worry). Questions are formulated as "how much of the time" or "how often have you experienced a problem," and a 1-7 Likert scale is used for the responses. The CLDQ-NAFLD has been adopted in the Chinese population with NAFLD.
Habitual Physical Activity and Dietary Intake | 16 weeks, 42 weeks
  The potential confounding factors in this project include habitual physical activity and dietary changes. We will control these factors by assessing them as outcome measures to be used as covariates in the data analyses to statistically control for potential confounding influences. We will thus measure the factors to monitor changes in physical activity and dietary intake over the study period. We are experienced in using actigraphy and the weighed food diary method to monitor and record habitual physical activity and diet.
Body Anthropometry-Waist circumference | 16 weeks, 42 weeks
  Waist circumference will be measured on bare skin midway between the lowest rib and superior border of the iliac crest using an inelastic measuring tape to the nearest 0.1 cm. Measurement will be performed at the end of normal expiration.

CONTACTS AND LOCATIONS:
Overall Officials: Parco M Siu, PhD, Principal Investigator — LKS Faculty of Medicine, The University of Hong Kong
Locations (1):
- LKS Faculty of Medicine, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The data of individual participants that underlie the results reported in this trial, after de-identification including text, tables, figures, and appendices, as well as study protocol and statistical analysis plan, will be shared after 3 months of study publication. Data will be shared with researchers who provide a methodologically sound proposal for academic purposes. Proposals should be directed to pmsiu@hku.hk to gain access and for data request, a data-access agreement needs to be signed.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 3 years following the publication of the article.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal for academic purposes. Proposals should be directed to pmsiu@hku.hk to gain access and for data request, a data-access agreement needs to be signed.